CLINICAL TRIAL: NCT00422123
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo Controlled, Phase III Study of the Efficacy and Safety of Quetiapine Fumarate (SEROQUEL®) Sustained-Release as Monotherapy in Adult Patients With Acute Bipolar Mania
Brief Title: Phase 3 /Seroquel SR Acute Mania Monotherapy - US
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D144CC00004
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Affective Psychosis, Bipolar; Manic Disorder; Manic-Depressive Psychosis; Mania; Manic State; Psychoses, Manic-Depressive
Keywords: Bipolar Disorder; Bipolar Mania; Manic Depression; Seroquel; Seroquel SR; quetiapine fumarate
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate (Seroquel) SR

SUMMARY:
The purpose of this study is to determine the safety and efficacy of sustained-release quetiapine fumarate (Seroquel®) in the treatment of patients with Acute Bipolar Mania for 3 weeks.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Documented diagnosis of Bipolar Disorder, with most recent episode being manic or mixed
* Inpatient hospital admission for the first 4 days of study treatment

Exclusion Criteria:

* >8 mood episodes within the last 12 months
* Use of prohibited medication
* Substance or alcohol abuse or dependence
* Current suicide risk or suicide attempt within last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2007-01; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to final visit in the YMRS total score

SECONDARY OUTCOMES:
Change from baseline to each visit in YMRS score and changes of YMRS subscores and changes in MADRS.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Datto, MD, Study Director — AstraZeneca; Larisa Acevedo, Ph.D, Study Director — AstraZeneca
Locations (51):
- United States (51):
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Cerritos, California
  - Research Site, Garden Grove, California
  - Research Site, Oceanside, California
  - Research Site, Pico Rivera, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Torrance, California
  - Research Site, Denver, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Aventura, Florida
  - Research Site, EAST Bradenton, Florida
  - Research Sitew, Fort Lauderdale, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, OAK Brook Terrace, Illinois
  - Research Site, Greenwood, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lake Charles, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Rockville, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Kenilworth, New Jersey
  - Research Site, Willingboro, New Jersey
  - Research Site, Elmsford, New York
  - Research Site, Holliswood, New York
  - Research Site, Durham, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Moon Township, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, DeSoto, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Arlington, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington

REFERENCES:
- [Derived] Cutler AJ, Datto C, Nordenhem A, Minkwitz M, Acevedo L, Darko D. Extended-release quetiapine as monotherapy for the treatment of adults with acute mania: a randomized, double-blind, 3-week trial. Clin Ther. 2011 Nov;33(11):1643-58. doi: 10.1016/j.clinthera.2011.10.002. Epub 2011 Nov 4. PMID 22054797